CLINICAL TRIAL: NCT07382232
Title: An RCT of Isometric Stability Versus Isotonic Mobility for LBP Rehabilitation
Brief Title: Isometric Stability vs. Isotonic Mobility for Chronic LBP
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palestine Ahliya University (Other)
Responsible Party: Principal Investigator, Azzam Alarab, Palestine Ahliya University is located in Jabal Daher, Bethlehem, West Bank, Palestine, with a mailing address of PO Box 1041, Bethlehem, ZIP code 90907, Palestine Ahliya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAUB
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: LBP
Keywords: Exercise therapy; LBP; Disability
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Group A: Isometric Exercises Group B: Isotonic Exercises
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm 1- Group A : Isometric Exercises (Experimental): • Isometric Exercise Group (IEG): This group performed a circuit of three core-stabilizing isometric exercises, each held for 10 seconds with brief rest intervals, for 5 complete repetitions. The exercises included: (a) Isometric Curl-Up, (b) Side Bridge, and (c) Bird Dog. The total dedicated exercise time was approximately 20 minutes per session.
  Interventions: Other: Isometric exercises
- arm2- Group B: Isotonic Exercises (Experimental): Isotonic Exercise Group (ITG): This group performed a circuit of three dynamic, strength-oriented isotonic exercises, each completed for 10 repetitions. The exercises included: (a) Bent Knee Sit-Up, (b) Cross Curl-Up, and (c) Prone Back Extension. The total dedicated exercise time was also approximately 20 minutes per session. All exercises were selected and adapted from previously published rehabilitation protocols for CLBP
  Interventions: Other: Isotonic exercises

INTERVENTIONS:
Other: Isometric exercises — • Isometric Exercise Group (IEG): This group performed a circuit of three core-stabilizing isometric exercises, each held for 10 seconds with brief rest intervals, for 5 complete repetitions. The exercises included: (a) Isometric Curl-Up, (b) Side Bridge, and (c) Bird Dog. The total dedicated exercise time was approximately 20 minutes per session.
  Arms: arm 1- Group A : Isometric Exercises
Other: Isotonic exercises — • Isotonic Exercise Group (ITG): This group performed a circuit of three dynamic, strength-oriented isotonic exercises, each completed for 10 repetitions. The exercises included: (a) Bent Knee Sit-Up, (b) Cross Curl-Up, and (c) Prone Back Extension. The total dedicated exercise time was also approximately 20 minutes per session. All exercises were selected and adapted from previously published rehabilitation protocols for CLBP [13].
  Arms: arm2- Group B: Isotonic Exercises

SUMMARY:
Background: Low back pain (LBP) is a leading cause of disability, often requiring primary care management.

Objective: To compare the effectiveness of isometric versus isotonic exercise programs for LBP.

Methods: Sixty adults with LBP were randomly assigned to two groups. Group A (n=30) performed isometric exercises, infrared therapy, and TENS. Group B (n=30) performed isotonic exercises with the same adjunct therapies. Pain (VAS), disability (MODI), and abdominal endurance were measured pre- and post-intervention.

Keywords: Exercise therapy; low back pain; disability evaluation

DETAILED DESCRIPTION:
Group-Specific Exercise Protocols:

* Isometric Exercise Group (IEG): This group performed a circuit of three core-stabilizing isometric exercises, each held for 10 seconds with brief rest intervals, for 5 complete repetitions. The exercises included: (a) Isometric Curl-Up, (b) Side Bridge, and (c) Bird Dog. The total dedicated exercise time was approximately 20 minutes per session.
* Isotonic Exercise Group (ITG): This group performed a circuit of three dynamic, strength-oriented isotonic exercises, each completed for 10 repetitions. The exercises included: (a) Bent Knee Sit-Up, (b) Cross Curl-Up, and (c) Prone Back Extension. The total dedicated exercise time was also approximately 20 minutes per session. All exercises were selected and adapted from previously published rehabilitation protocols for CLBP [13].

Adjunctive Therapies (Common to Both Groups):

1. Infrared (IR) Therapy: A standard therapeutic infrared lamp was positioned 50 cm from the participant's lumbar spine at a 90-degree angle. Heat was applied for 15 minutes per session to promote muscle relaxation and local blood flow.
2. Transcutaneous Electrical Nerve Stimulation (TENS): Electrodes were placed over the painful lumbar area. A low-frequency (<10 Hz) TENS unit was applied for 20 minutes per session. The analgesic mechanism of TENS is well-documented, involving the modulation of pain pathways via opioid and noradrenergic receptors in the central nervous system [16].

Both groups received a standardized four-week intervention program, consisting of three supervised sessions per week, totaling 12 sessions. Each 55-minute session included adjunctive therapies common to both groups, followed by the specific exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years;
* Diagnosis of non-specific CLBP, defined as pain localized between the lower rib margin and the gluteal folds persisting for more than three months;
* Self-reported pain intensity score between 40 mm and 80 mm on a 100-mm Visual Analogue Scale (VAS), indicating moderate to severe pain;
* Pain experienced on at least three days in the month preceding enrollment, with documented interference in daily activities;
* A formal referral for physiotherapy management.

Exclusion Criteria:

* The presence of "red flag" pathologies (e.g., spinal tumor, infection, fracture); - Neurological signs or symptoms suggestive of radiculopathy or myelopathy;
* a history of spinal surgery or epidural steroid injections within the previous 12 months;
* Systemic inflammatory diseases (e.g., rheumatoid arthritis) or major neurological disorders;
* Pregnancy;
* Receipt of physiotherapy for low back pain within the last six months;
* Current use of non-steroidal anti-inflammatory drugs (NSAIDs) or inability to refrain from their use during the study period;
* Any diagnosed psychiatric condition.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
VAS | 4 WEEKS
  Measured using a 100-mm Visual Analogue Scale , where 0 mm represents "no pain" and 100 mm represents "the worst pain imaginable." Participants marked a point on the line corresponding to their current pain level. The Arabic version of the VAS has been validated as a reliable and responsive tool for pain assessment in clinical populations [17].

SECONDARY OUTCOMES:
MODI | 4WEEKS
  This self-administered questionnaire contains 10 items addressing various aspects of daily life (e.g., pain intensity, personal care, lifting, walking). Each item is scored from 0 to 5, with the total sum converted to a percentage (0-100%); higher scores indicate greater disability. The MODI is a gold-standard tool with demonstrated high reliability, validity, and sensitivity to clinical change in patients with low back pain [18].
Muscular Endurance | 4WWEKS
  Assessed via a standardized Abdominal Endurance Test. Participants were instructed to hold a partial curl-up position (trunk elevated at 30° from the plinth) for as long as possible while maintaining proper form. The time in seconds until failure was recorded. This test is a validated and reliable measure of core muscular endurance, a key component of lumbar stability [19].

CONTACTS AND LOCATIONS:
Locations (1):
- Palestine Ahliya University, Bethlehem, West Bank, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No